CLINICAL TRIAL: NCT05817981
Title: The Investigation of Knowledge, Attitude/Belief, Practice (KAP) and Educational Demand Analysis of Sexual and Reproductive Health Among Adolescent and Young Adult Cancer Survivors in the Context of Healthy China
Brief Title: The Investigation of Knowledge and Educational Demand of Sexual and Reproductive Health Among Cancer Survivors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wei XIA, PhD, Philosophic Doctor, Sun Yat-sen University
Other Study IDs: pdjh2023 b0020
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Sexual and Reproductive Health
Keywords: sexual and reproductive health; adolescent and young adult; knowledge，attitude/belief，practice; educational demand
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adolescent and Young Adult Cancer Survivors: Adolescent and young adult cancer survivors who aged range from 15 to 39, having been diagnosed with cancer and completed cancer treatment for at least 6 months.
  Interventions: Other: Semi-structured interview; Other: Questionnaires set
- Clinical oncology medical staff: Medical staff who routinely work in the oncology ward.
  Interventions: Other: Semi-structured interview

INTERVENTIONS:
Other: Semi-structured interview — Before the questionnaire survey, 30 cancer survivors and 30 clinical oncology medical staff will respectively participate in different semi-structured interview individually.
Other: Questionnaires set — Except for participants who participated in semi-structured interviews, other cancer survivors who met the inclusion criteria will be asked to respond to the demographic information sheet, the cancer related sexual and reproductive health knowledge and attitudes questionnaire, and the access methods and demand for cancer-related fertility information.
  Groups: Adolescent and Young Adult Cancer Survivors

SUMMARY:
The goal of this observational study is to explore the current situation and needs of adolescent and young adult cancer survivors for cancer-related reproductive health and fertility information. The main questions it aims to answer are:

1. What is the status of sexual and reproductive health knowledge among adolescent and young adult cancer survivors?
2. What is the difference between the educational currently available and needs of cancer survivors? Part of the participants will be interviewed and then others will fill out questionnaires.

DETAILED DESCRIPTION:
Cancer is a major public health problem worldwide. With the development of medical and diagnostic technology, the number of cancer survivors worldwide continues to grow, especially among adolescents and young adults. The global average cure rate for pediatric cancer patients was 52%, and the 5-year survival rates of this population in developed countries were about 80% in recent years. With this trend, more pediatric cancer patients are transitioning into the ranks of adolescent cancer survivors.

The fertility intention is generally strong among adolescent and young adult cancer survivors, more than three quarters of non-fertile cancer survivors have a high desire to have children. However, most of them have an unfulfilled desire to have their own child, which lead to high levels of fertility anxiety. What's more, studies have shown that adolescent and young adult cancer survivors also have a great need for sexual and reproductive health, but relevant forms of health care are rarely existed. Young and adolescent cancer survivors are limited by the age of illness and generally lack regular sexual and reproductive health education in schools. Due to the long and painful cancer treatments, they also have difficulty in obtaining relevant knowledge or reproductive health education from professionals such as doctors or nurses during cancer treatment. The lack of communication between providers of survival care services and between providers and survivors makes the sexual and reproductive health education much more difficult for cancer survivors. Numerous studies have shown that a lack of knowledge about reproductive health leads to increased psychological burden, low quality of life and depression among young cancer survivors. Thus, it is critical to meet the reproductive health literacy needs of young people and adolescent cancer survivors.

China is in the midst of an era of optimized birth and three-child policy, but the fertility policy for cancer survivors is relatively poor. Survival care in China currently focuses on the monitoring, prevention and treatment of delayed physical and mental reactions caused by cancer itself and its treatment in adolescent and young adult cancer survivors. Health promotion, such as sexual and reproductive health, or quality of life for survivors is rarely discussed. To some extent, high-quality, multichannel reproductive health counseling and health education may alleviate fertility concerns for adolescent and young adult cancer survivors and improve long-term quality of life. Therefore, on the basis of continuing to provide long-term care for adolescent and young adult cancer survivors, it is necessary to increase sexual and reproductive health counseling, health education and other services for this population. What's more, providing sexual and reproductive health related knowledge through multiple channels can improve the long-term quality of life for adolescents and adolescents.

Before applying interventions to help adolescent and young adult cancer survivors to access to cancer-related reproductive health information, a study exploring their intention to acquire knowledge and relevant factors must be implemented.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent and young adult cancer survivors: ①be aged range from 15 to 39, ②have been diagnosed with cancer and completed cancer treatment for at least 6 months, ③be able to read, understand and communicate in Chinese.
* Clinical oncology medical staff: ①are clinician or nurse specialist in oncology, ②the average daily contact time with patients in clinical work is not less than 20% of the clinical working time.

Exclusion Criteria:

* Adolescent and young adult cancer survivors: ①unable to complete communication due to serious mental or physical illness such as deaf-mute, mental illness resulting in unclear consciousness, ②be cancer recurrence or second cancer at screening.

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The NCCS defined someone as a cancer survivor from the moment of diagnosis through to the end of life.
Sampling Method: Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Knowledge and attitudes about sexual and reproductive health related to cancer | Baseline
  According to the qualitative research results and literature review, the questionnaire items can be tentatively prepared to cover the impact of cancer itself and the impact of treatment methods (such as surgery, radiotherapy, chemotherapy, hormone therapy, etc.) on reproductive function, the survivors' own reproductive function impairment, pregnancy risk, pregnancy risk, etc. Using the Likert level 5 scoring method, based on the level of the answer of each item,1 point means "completely unclear" and 5 points means "very clear".

SECONDARY OUTCOMES:
Socio-demographic information | Baseline
  The socio-demographic data collected through the structural questionnaire includes gender, age, family income, personal education level, marital status, fertility status, parents' education level, family income; cancer type, diagnosis time, completed treatment, medication, treatment completion time and completion degree.
Access methods and demand for cancer-related fertility information | Baseline
  Referring to the questionnaire designed by B. Elizabeth Oosterhuis's research team, combined with the qualitative research results and China's national conditions, we have preliminarily formulated six options: oncologists, responsible nurses, doctors specializing in reproductive medicine, information materials distributed by hospitals, conversations with other cancer patients and through the website/Internet.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xia, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No